CLINICAL TRIAL: NCT00397475
Title: Evaluation of Colecalciferol Substitution in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 142/06
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: RENAL INSUFFICIENCY, CHRONIC; Hyperparathyroidism, Secondary
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cholecalciferol

INTERVENTIONS:
Drug: Colecalciferol

SUMMARY:
The purpose of this study is to determine the effect of a colecalciferol substitution in dialysis patients on bone metabolism and immune system

ELIGIBILITY:
Inclusion Criteria:

1. Serum 25-OH-Vit.D-levels < 60 ng/ml
2. Age > 18 years
3. dialysis treatment > 3 Months
4. signed written informed consent
5. Serum-Calcium-levels < 2,6 mmol/l within the last 4 weeks
6. Serum-Phosphate-levels < 7,0 mg/dl within the last 4 weeks
7. Ca x P-Product < 75 mg2/dl2 within the last 4 weeks

Exclusion Criteria:

1. Serum 25-OH-Vit.-D-levels > 60 ng/ml
2. concommitant participation in another interventional trial
3. psychiatric disorders preventing from valid informed consent
4. Hyperphosphatemia (> 7,0 mg/dl) within the last 4 weeks
5. Hypercalcemia (> 2,6 mmol/l) within the last 4 weeks
6. Ca x P-Product > 75 mg2/dl2 within the last 4 weeks
7. pregnancy or lactation
8. known malignancy
9. liver disease, defined as 2-fold upper limit of ASAT-, or ALAT-levels
10. PTH levels < 50 pg/ml
11. current clinically relevant infections treated with antibiotic therapy and raised hsCRP levels
12. Chronic viral Infectious diseases (e.g. HIV, Hepatitis B or C)
13. Immunosuppressant Medication
14. known hematologic disorders, other than renal anemia
15. age below 18 years
16. known anaphylactic reaction against the study medication or other ingredients of the study drug preparation
17. renal calculus
18. Pseudohypoparathyroidism
19. Medication including cardiac glycosides
20. Sarkoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
CD14/CD16-Monocyte-Subsets (Frequency)

SECONDARY OUTCOMES:
Production of Cytokines: IFN-γ, TNF-α
Serum levels of Calcium, Phosphorus, iPTH, hsCRP, alkaline phosphatase
Th1/Th2- and Tc1/Tc2-Lymphocyte-Frequency

CONTACTS AND LOCATIONS:
Overall Officials: Eric Seibert, M.D., Principal Investigator — University Hospital of Saarland, Dpt. of Internal Medicine IV, Div. of Nephrology and Hypertension
Locations (1):
- University Hospital of Saarland, Dpt. of Internal Medicine IV, Div. of Nephrology and Hypertension, Homburg, Saarland, Germany